CLINICAL TRIAL: NCT05911256
Title: TEAM Support to Improve Glycemic Control Using CGM in Diverse Populations
Brief Title: A Community Health Worker/Pharmacist Team to Improve Blood Sugars in Diabetes Care Using Continuous Glucose Monitoring
Acronym: TEAM-CGM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Baystate Health (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ben Gerber, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000848; R01DK133265 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pharmacist Only (Active Comparator): Participants will receive clinical pharmacist management of diabetes. Those participants who meet their HbA1c goal at 6 months will continue with maintenance diabetes management. This includes routine primary care with the primary care provider, routine medication management, and traditional home glucose monitoring. For those not meeting goals in HbA1c they will be randomized again to receive Pharmacist + CGM or receive Pharmacist + CGM + Community Health Worker (CHW) support.
  Interventions: Behavioral: Pharmacist Only
- Pharmacist + CGM (Experimental): Participants receive clinical pharmacist + CGM support. Those participants who meet their HbA1c goal at 6-months will continue with maintenance diabetes management. This includes routine primary care with the primary care provider, routine medication management, and traditional home glucose monitoring. For those not meeting goals in HbA1c, they will be randomized again to continue with pharmacist + CGM or receive additional CHW support (Pharmacist + CGM + CHW).
  Interventions: Behavioral: Pharmacist Only; Device: Continuous Glucose Monitor (CGM)
- Pharmacist + CGM + CHW (Experimental): A second randomization step occurs at 6-months. Participants randomized to this condition receive clinical pharmacist, CHW, and CGM support.
  Interventions: Behavioral: Pharmacist Only; Device: Continuous Glucose Monitor (CGM); Behavioral: Community Health Worker (CHW)

INTERVENTIONS:
Behavioral: Pharmacist Only — Clinical pharmacists conduct encounters with patients by videoconferencing or phone. Pharmacists conduct a broad range of activities including ongoing evaluation of medication and lifestyle adherence, setting therapeutic goals, formulating a provider-approved plan of care, and documenting the plan in the electronic health record. Pharmacists propose medication changes based on algorithms and protocols derived from national guidelines under physician guidance.
Device: Continuous Glucose Monitor (CGM) — Patients will receive the Continuous Glucose Monitoring (CGM) system. The instruction on use of device is the intervention being tested, not the effectiveness of the device itself. Participants will receive instruction and training on how to use the device and will wear the device for 10 days.
  Arms: Pharmacist + CGM; Pharmacist + CGM + CHW
Behavioral: Community Health Worker (CHW) — Patients are connected to a community health worker(CHW). CHWs conduct home visits and facilitate 3-way Telehealth visits (Patients, pharmacists, and CHWs) via an iPad with cellular plan. Additional CHW activities include social determinants of health screening, health behavior education, problem solving, goal setting, and medication adherence support.
  Arms: Pharmacist + CGM + CHW

SUMMARY:
Continuous glucose monitoring (CGM) can help improve blood sugar management in type 2 diabetes. A sequential, multiple assignment, randomized trial will evaluate clinical pharmacists, community health workers, and telehealth in supporting CGM use to improve blood sugar control.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) has demonstrable benefits for people living with diabetes, including improvement in diabetes control and reduction in hypoglycemia. Randomized controlled trials have demonstrated that CGM can reduce hemoglobin A1c (HbA1c) and increase in the time in range metric. Little is known about CGM use in the broader population with type 2 diabetes (T2DM) in low-income, minority populations not receiving insulin therapy. This proposed study will rigorously evaluate CGM in a diverse and vulnerable population with T2DM in the primary care setting. The proposed study will integrate CGM into the study team's previously studied approach of mobile health (mHealth) diabetes management. The investigators prior research has leveraged mHealth tools and a community health worker (CHW)/clinical pharmacist team to manage low-income, minority populations with T2DM. Clinical pharmacists embedded in the healthcare system review patient glucose levels, promote medication adherence and collaboratively adjust therapy to help patients reach HbA1c goals. CHWs augment pharmacist-led efforts and address social determinants of health and provide individualized, contextual self-management support. In partnership with Baystate Community Health Centers and UMass Memorial Health, the investigators propose an effectiveness study of team-supported CGM using a Sequential Multiple Assignment Randomized Trial (SMART) study design. The investigators plan to study a diverse population with 318 T2DM patients receiving pharmacist- and CHW-supported CGM delivered through community health centers in Massachusetts. The Specific Aims include: (1) Conduct a randomized, controlled trial to evaluate the effectiveness of pharmacist-supported CGM in a diverse patient population with T2DM in the primary care setting. The investigators hypothesize that pharmacist-supported CGM will result in improved HbA1c, CGM metrics, and other secondary outcomes (e.g., quality of life) at 6 months compared with pharmacist-only care; (2) Re-randomize patients not at HbA1c goal after 6 months to receive or not receive CHW support beyond pharmacist-supported CGM. The investigators hypothesize that adding CHWs will result in improved HbA1c, CGM metrics, and other secondary outcomes at 12 months compared with pharmacist-supported CGM alone; (3) Evaluate reach, effectiveness, adoption, implementation, and maintenance using the RE-AIM framework; and (4) Determine total cost and cost-effectiveness of CGM and the supportive components (e.g., clinical pharmacist and CHW) from the perspective of the healthcare organization. If this team support model of diabetes care is found to be cost-effective, such evidence may influence insurance restrictions on ambulatory CGM coverage in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-75.
* History of T2DM > 1 year.
* Speak English or Spanish.
* A1c ≥ 8% (within past 6 months) - with reduction if necessary based on recruitment.
* eGFR (estimated glomerular filtration rate) > 30.
* Willingness to use continuous glucose monitoring (CGM) and work with a community health worker (including home visits) and clinical pharmacist.

Exclusion Criteria:

* Plans for weight reduction surgery or prescription weight loss medication (specific for weight loss, not GLP-1).
* Current, recent, or planned use of CGM.
* Current use of steroids.
* Abuse of illicit drugs.
* Pregnancy (or planned pregnancy).
* Specific comorbidities (e.g., recent MI, TIA, CVA, malignancy, hemoglobinopathy, severe hypoglycemia, etc.).
* Psychiatric disorder that may limit ability to perform study tasks
* Skin changes that preclude use of sensor or allergy to adhesive.
* Planning to leave geographic area within 12 months or distance from clinical site > 20 miles.
* Participation in another study.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in participant HbA1c values | 0, 3, 6, 9, and 12 months (and additional 18-month collection in first 75% of participants)
  Participant HbA1c will be measured and obtained by finger stick using home testing kits.

SECONDARY OUTCOMES:
Change in glycemic control from baseline using Percent Time in Range | 0, 6, and 12 months
  The percentage of time when blood glucose was between 70 and 180 mg/dl, percentage of time when blood glucose was greater than 250mg/dL , and percentage of time when glucose was les than 70mg/dL. as measured by the continuous glucose monitor
Change in Participant self-reported health-related quality of life from baseline | 0, 6, and 12 months
  Participant self-reported health related quality of life will be measured using EQ-5D (not an abbreviation), a standardized measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health. 1)Mobility, 2)Self-Care 3) Usual Activities 4)Pain and Discomfort 5)Anxiety and Depression. 'Scores for each dimension range from 1-3 with higher scores indicating lower quality/worse outcomes
Change in participant reported Diabetes Self-Management from baseline | 0, 6, and 12 months
  Diabetes Self-Management will be measured using Diabetes Self-Management Questionnaire (DSMQ) is a 16 item questionnaire use to assess self-care activities associated with glycemic control. Scores range from 0 to 10 with higher scores associated with poorer diabetes self-management.
Changes in participant reported Diabetes Distress from baseline | 0, 6, and 12 months
  Participant reported Diabetes Distress will be measured using the Diabetes Distress Scale (DDS) is a 17 -item scale that captures you critical dimensions of distress for individuals with Diabetes: emotional burden, regimen distress, interpersonal distress, and physician distress. The DDS results in an overall distress score ranging from 1 to 6 with higher scores indicating greater distress. The DDS also yields 4 sub scale scores for each 4 dimensions of distress with scores ranging from 1 to 6, with higher scores indicating greater distress.
Change in participant-reported diabetes treatment burden from baseline | 0, 6, and 12 months
  Participant reported diabetes treatment burden will be assessed using the Diabetes Treatment Burden Questionnaire(DTBQ). The DTBQ is an 18-item questionnaire that assesses the treatment burden caused by pharmacotherapy for type 2 diabetes. Scores range from 0 to 6 with 0 corresponding to minimum burden, and 6 corresponding to maximum burden.
Frequency of participant Healthcare Utilization | 0, 6, and 12 months
  Participant Healthcare utilization will be measured with a 3-question survey to capture the frequency of Emergency Room visits, calls to 911, after hours/urgent care visits, and dietician visits. This survey includes encounters whether diabetes-related or not.
Change in mean glycemic control from baseline | 0,6,12 months
  Mean glucose as measured by the continuous glucose monitor
Hyperglycemia event rate | 0, 6, 12 months
  Number of hyperglycemic events as measured by the continuous glucose monitor
Change in Glycemic variability from baseline | 0, 6, 12 months
  This will be measured by the continuous glucose monitor, the coefficient of variation in glucose variability will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Gerber, MD, MPH, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant survey data, participant physiologic data, community health worker training and protocol, clinical pharmacist training and protocol, will be shared. This includes a complete, de-identified data set, including survey and clinical/physiologic data (and relevant R or SAS code) through DKnet, the Inter-University Consortium for Political and Social Research, or eScholarship@UMassChan.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will become available at time of primary results publication.